CLINICAL TRIAL: NCT02182648
Title: Bispectral Index Guiding Etomidate Used in Children Aged 3 to 10 for Clinical Anesthesia Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: etomidate children 20140625
Record Dates: First submitted 2014-06-29; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Bispectral Index; Pediatric; Etomidate; Induction
MeSH Terms: interventions — Etomidate; Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- etomidate group (Experimental): infusion of etomidate at 2 minutes before anesthesia induction
  Interventions: Drug: etomidate
- propofol group (Active Comparator): infusion of propofol at 2 minutes before anesthesia induction
  Interventions: Drug: propofol
- sevoflurane group (Active Comparator): inhale sevoflurane for anesthesia induction and maintenance
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: etomidate — 1. intravenous injection midazolam 0.08 mg/kg, fentanyl 0.002 mg/kg, cisatracurium 0.15 mg/kg for induction of anesthesia.
  2. infusion of etomidate at 2 minutes before anesthesia induction
  Arms: etomidate group
Drug: propofol — 1. intravenous injection midazolam 0.08 mg/kg, fentanyl 0.002 mg/kg, cisatracurium 0.15 mg/kg for induction of anesthesia.
  2. infusion of propofol at 2 minutes before anesthesia induction
  Arms: propofol group
Drug: sevoflurane — 1. intravenous injection midazolam 0.08 mg/kg, fentanyl 0.002 mg/kg, cisatracurium 0.15 mg/kg for induction of anesthesia.
  2. inhale sevoflurane for anesthesia induction and maintenance
  Arms: sevoflurane group

SUMMARY:
This research through using bispectral index to guide the induced dose and speed of etomidate lipid emulsion for pediatric total venous anesthesia,and to provide a reference for clinical anesthesia physician.

ELIGIBILITY:
Inclusion Criteria:

1. obtain informed consent;
2. undergoing elective hypospadias repair surgery under general anesthesia;
3. American society of anesthesiologists (ASA) class I-II;
4. aged between 3-10 years old;
5. BMI is 18.5-30 kg/m2;

Exclusion Criteria:

1. systolic blood pressure≥180 mmHg or<90 mmHg, diastolic blood pressure≥110 mmHg or<60 mmHg;
2. serious heart, brain, liver, kidney, lung, endocrine diseases or serious infections;
3. long-term use of hormone or a history of adrenal cortex inhibition;
4. suspected or confirmed difficult airway;
5. suspected or confirmed abuse of narcotic analgesic drugs, psychotropic drugs;
6. neuromuscular disease;
7. mental instability, or have a mental illness;
8. allergic to investigational products or with other contraindication
9. participated in other study within 30 days

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
the amount of drugs | from the beginning of induction to Bispectral Index < 50,up to 5 minutes
  the amount of etomidate,propofol and sevoflurane used in anesthesia induction
the drugs used time | from the beginning of induction to Bispectral Index < 50,expected to be within 1 minute
  the injection time of etomidate and propofol, and the inhale time of sevoflurane during anesthesia induction
numbers of muscular fibrillation | from the beginning of induction to Bispectral Index < 50,up to 5 minutes
  numbers of muscular fibrillation in anesthesia induction
degree of inflammation reaction | baseline,5 minutes after indution,5 minutes before operation end,30 mimutes、24h and 48h after operation
  serum levels of interleukin 6 and tumor necrosis factor α will be measured at each time point using ELISA method
adrenal function | baseline,5 minutes after indution,5 minutes before operation end,30 mimutes、24h and 48h after operation
  serum level of cortisol will be measured at each time point using radioimmunoassay

SECONDARY OUTCOMES:
hemodynamic parameters | from the beginning of induction to skin closure, up to 3 hours
  heart rate,blood pressure,electrocardiogram and pulse oxygen saturation recorded at 4 time points including before anesthesia induction,before endotracheal intubation,after endotracheal intubation and after operation immediately
sedation degree | from the beginning of induction to skin closure, up to 3 hours
  Bispectral index,train-of-four stimulation and the temperature recorded at 4 time points including before anesthesia induction,before endotracheal intubation,after endotracheal intubation and after operation immediately